CLINICAL TRIAL: NCT00685945
Title: Renin-Angiotensin Aldosterone System and Fibrinolysis(RAAS) Interaction in Humans- Specific Aim 3
Brief Title: Renin-Angiotensin Aldosterone System and Fibrinolysis Interaction in Humans-Specific Aim 3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Center for Research Resources (NCRR) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Nancy J. Brown, Professor of Medicine and Clinical Pharmacology, Vanderbilt University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Health Services Research
Other Study IDs: RAAS & Fibrinolysis; 2R01HL060906 (NIH); HL065193 (Other Grant/Funding Number: NIH); UL1RR024975 (NIH); 5R01HL085740-05 (NIH)
Record Dates: First submitted 2008-05-27; First posted 2008-05-29 (Estimated); Results first posted 2013-02-25 (Estimated); Last update posted 2013-02-25 (Estimated); Status verified 2013-01

CONDITIONS: Obesity
Keywords: Bradykinin; Obesity; Nitric Oxide Donor; tissue type plasminogen activator; isosorbide dinitrate; phosphodiesterase inhibitor; Renin-Angiotensin Aldosterone System; Fibrinolysis; Angiotensin converting enzyme
MeSH Terms: conditions — Obesity | interventions — Bradykinin; omega-N-Methylarginine; Isosorbide; Sildenafil Citrate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Control (bradykinin infusion) (Experimental): Bradykinin (Clinalfa AG, Läufelfingen, Switzerland)
  Interventions: Drug: Control (bradykinin)
- L-NMMA + bradykinin (Experimental): N-monomethyl-L-arginine (L-NMMA, NO synthase inhibitor; Bachem, Torrance, CA)
  Interventions: Drug: L-NMMA + bradykinin
- Isosorbide + L-NMMA + bradykinin (Experimental): Isosorbide (NO donor)
  Interventions: Drug: Isosorbide + L-NMMA + bradykinin
- Sildenafil + L-NMMA + bradykinin (Experimental): Sildenafil (phosphodiesterase type 5 (PDE5) inhibitor
  Interventions: Drug: Sildenafil + L-NMMA + bradykinin

INTERVENTIONS:
Drug: Control (bradykinin) — Graded doses of bradykinin (Clinalfa AG, Läufelfingen, Switzerland) will be infused at 50, 100, and 200ng/min. Each dose will be infused for 5 minutes and FBF will measured during the last 2 minutes of infusion. Arterial and venous blood samples will be obtained for measurement of net t-PA release after each dose.
  Arms: Control (bradykinin infusion)
Drug: L-NMMA + bradykinin — Thirty minutes after administration of bradykinin a continuous intra-arterial infusion of L-NMMA at 12 micromol/min will be started started. While continuing the infusion of L-NMMA, baseline measurements and infusion of bradykinin will be repeated.
  Other Names: N-monomethyl-L-arginine
  Arms: L-NMMA + bradykinin
Drug: Isosorbide + L-NMMA + bradykinin — Following the second bradykinin infusion, 12 subjects will receive 5mg isosorbide dinitrate (an exogenous NO donor; Major Pharmaceuticals Inc, Livonia MI). Sixty minutes after the administration of isosorbide the continuous intra-arterial infusion of L-NMMA at 12 micromol/min will be restarted and baseline measurements and bradykinin infusion will be repeated.
  Arms: Isosorbide + L-NMMA + bradykinin
Drug: Sildenafil + L-NMMA + bradykinin — Following the second bradykinin infusion, 12 subjects will receive 50mg sildenafil (phosphodiesterase type 5 (PDE5) inhibitor to increase cGMP without increasing NO; Pfizer, NY). Sixty minutes after the administration of sildenafil the continuous intra-arterial infusion of L-NMMA at 12 micromol/min will be restarted and baseline measurements and bradykinin infusion will be repeated.
  Arms: Sildenafil + L-NMMA + bradykinin

SUMMARY:
The purpose of the study is to determine if giving isosorbide,a drug that is used to treat chest pain, affects blood vessel release of an anti-clotting factor.

DETAILED DESCRIPTION:
To test the hypothesis that the administration of the NO donor isosorbide dinitrate,but not the phosphodiesterase inhibitor sildenafil, will attenuate stimulated vascular t-PA release whereas both agents will improve glucose uptake.

ELIGIBILITY:
Inclusion Criteria:

* 18-70 years of age
* Male and female subjects
* Surgical sterilization
* Childbearing potential: beta HCG on study day
* Subjects with a body mass index of 25 or greater

Exclusion Criteria:

* Diabetes type 1 to type 2 as defined by a fasting glucose of 126 mg/dl or greater or the use of anti-diabetic medication
* Use of hormone replacement therapy
* Statin therapy
* In hypertensive subjects, a seated systolic blood pressure greater than 179 mmHg or a seated diastolic blood pressure greater than 110 mmHg or taking hypertensives
* Pregnancy/Breast Feeding
* Cardiovascular disease such as myocardial infarction with 6 months prior to enrollment, presence of angina pectoris, significant arrhythmia, congestive heart failure (LV hypertrophy acceptable) deep vein thrombosis, pulmonary embolism, second or three degree heart block, mitral valve stenosis, aortic stenosis, or hypertrophic cardiomyopathy
* Treatment with anticoagulants
* History of serious neurologic disease such as cerebral hemorrhage, stroke or transient ischemic attack
* Diagnosis of asthma
* Clinically significant gastrointestinal impairment that could interfere with drug absorption
* Hematocrit <35%
* Hyperlipidemic fasting Total Cholesterol >220mg/dl
* Impaired renal function (Serum creatinine >1.5 mg/dl)
* History or presence of immunological or hematological disorders
* Any underlying or acute disease requiring regular medication which could possible pose a threat to the subject or make implementation of the protocol or interpretation of the study results difficult
* Impaired hepatic function (Serum glutamic oxaloacetic transaminase, serum glutamate pyruvate transaminase > 60)
* Treatment with chronic systemic glucocorticoid therapy (more than 7 days in 1 month)
* Treatment with lithium salts
* History of Alcohol or drug abuse
* Treatment with any investigational drug 1 month preceding study
* Mental conditions rendering the subject unable to understand the nature, scope and possible consequences of the study
* Inability to comply with the protocol

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2007-12; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nancy J Brown, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center-GCRC, Nashville, Tennessee, United States

REFERENCES:
- [Result] Pretorius M, Brown NJ. Endogenous nitric oxide contributes to bradykinin-stimulated glucose uptake but attenuates vascular tissue-type plasminogen activator release. J Pharmacol Exp Ther. 2010 Jan;332(1):291-7. doi: 10.1124/jpet.109.160168. Epub 2009 Oct 19. PMID 19841473

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from a volunteer registry at Vanderbilt University. Subjects who participated in prior studies and requested to be contacted for future studies were included in the recruitment process. Recruitment began on 12/07 and stopped on 1/09.
Pre-assignment Details: Subjects with renal, endocrine, hematological or cardiovascular disease (including hypertension defined as an untreated systolic/diastolic blood pressure greater than 140/90 mmHg were excluded. Subjects with a fasting cholesterol greater than 5.7 mmol/L (220 mg/dl) and smokers were excluded. No washout period was required for the study.
Groups:
- All Participants: 24 subjects received a bradykinin infusion and then a bradykinin + L-NMMA infusion. Subjects were then randomized to receive either isosorbide (N=12) or sildenafil (N=12). The infusion of bradykinin + L-NMMA was then repeated.
Period: Control (Bradykinin Infusion)
Arm/Group | All Participants
Started | 24 (A total of 24 subjects received an infusion of bradykinin)
Completed | 24
Not Completed | 0
Period: L-NMMA + Bradykinin
Arm/Group | All Participants
Started | 24
Completed | 23
Not Completed | 1
Not completed — Physician Decision | 1
Period: Isosorbide + L-NMMA + Bradykinin
Arm/Group | All Participants
Started | 11
Completed | 11
Not Completed | 0
Period: Sildenafil + L-NMMA + Bradykinin
Arm/Group | All Participants
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: Subjects characteristics for all 24 participants
Arm/Group | All Participants
Number analyzed (Participants) | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 24
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 31.71 (6.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 12
Region of Enrollment [Number; unit: participants]
  United States | 24

OUTCOME MEASURES:

1. Primary Outcome: Net Tissue-type Plasminogen Activator (t-PA) Release
Description: Individual net t-PA release at each time point were calculated by the following formula: net release = (Cv-CA) x {FBF x [101-hematocrit/100]}, where Cv and CA represent the concentration of t-PA in the brachial vein and artery, respectively.
Time Frame: During and after each study drug administration
Population: Twenty four subjects were studied. One subject was excluded because of erroneous drug administration. Analysis was per protocol. Twenty-three subjects receive bradykinin then L-NMMA plus bradykinin infusions. Subjects were then randomized to either isosorbide or sildenafil. Twelve subjects received sildenafil and 11 subjects received isosorbide.
Measure: Mean (Standard Error); unit: ng/min/100ml
Groups:
- Control: Subjects received bradykinin at 50, 100 and 200ng/min
- L-NMMA + Control: After the intial bradykinin infusion subjects then received a continuous infusion of L-NMMA plus bradykinin at 50, 100 and 200ng/min
- Isosorbide + L-NMMA + Control: Eleven of the twenty-four subjects were randomized to isosorbide after completing the bradykinin and bradykinin plus L-NMMA infusions. The bradykinin plus L-NMMA infusions were then repeated.
- Sildenafil + L-NMMA + Control: Twelve of the twenty-four subjects were randomized to sildenafil after completing the bradykinin and bradykinin plus L-NMMA infusions. After 1 hour, bradykinin plus L-NMMA infusions were repeated.
Arm/Group | Control | L-NMMA + Control | Isosorbide + L-NMMA + Control | Sildenafil + L-NMMA + Control
Number analyzed (Participants) | 24 | 23 | 11 | 12
ng/min/100ml
  Net t-PA release (bradykinin 0ng/min) | 0.24 (0.39) | 0.59 (0.23) | -0.38 (0.51) | 0.29 (0.67)
  Net t-PA release (bradykinin 50ng/min) | 1.02 (1.06) | 3.65 (0.79) | 3.14 (1.13) | 2.46 (2.07)
  Net t-PA release (bradykinin 100ng/min) | 11.81 (2.12) | 22.10 (5.51) | 15.90 (3.13) | 18.48 (9.11)
  Net t-PA release (bradykinin 200ng/min) | 30.03 (4.24) | 39.90 (6.98) | 45.32 (9.45) | 37.39 (11.79)
Statistical Analysis 1: Comparison: Control vs L-NMMA + Control vs Isosorbide + L-NMMA + Control vs Sildenafil + L-NMMA + Control; The effect of bradykinin on net t-PA release was determined using general linear model-repeated measures ANOVA in which the between-subject variable was gender, and the within-subjects variables were drug (control, +L-NMMA, +L-NMMA plus isosorbide, or +L-NMMA plus sildenafil) and dose of bradykinin; Test type: Superiority or Other; p = 0.04, ANOVA

2. Secondary Outcome: Forearm Blood Flow (FBF)
Description: Forearm blood flow was measured by strain gauge plethysmography
Time Frame: During and after each study drug administration
Measure: Mean (Standard Error); unit: ml/min/100ml
Groups:
- L-NMMA + Control: Subjects received a continuous infusion of L-NMMA plus bradykinin at 50, 100 and 200ng/min
- Isosorbide + L-NMMA + Control: Twelve (of the twenty-four)subjects received isosorbide after completing the bradykinin and bradykinin plus L-NMMA infusions. The bradykinin plus L-NMMA infusions were then repeated.
- Sildenafil + L-NMMA + Control: Twelve (of the twenty-four) subjects received sildenafil after completing the bradykinin and bradykinin plus L-NMMA infusions. After 1 hour, bradykinin plus L-NMMA infusions were repeated.
Arm/Group | Control | L-NMMA + Control | Isosorbide + L-NMMA + Control | Sildenafil + L-NMMA + Control
Number analyzed (Participants) | 24 | 23 | 11 | 12
ml/min/100ml
  FBF (bradykinin 0 ng/min) | 4.03 (0.25) | 2.36 (0.18) | 2.18 (0.33) | 2.80 (0.37)
  FBF (bradykinin 50ng/min) | 7.02 (0.57) | 5.16 (0.37) | 4.73 (0.70) | 5.87 (0.79)
  FBF (bradykinin 100ng/min) | 13.17 (1.04) | 8.67 (0.81) | 6.83 (1.13) | 9.13 (0.76)
  FBF (bradykinin 200 ng/min) | 17.74 (1.43) | 11.21 (1.12) | 9.91 (1.72) | 12.92 (1.30)
Statistical Analysis 1: Comparison: Control vs L-NMMA + Control vs Isosorbide + L-NMMA + Control vs Sildenafil + L-NMMA + Control; Test type: Superiority or Other; p < 0.001, ANOVA; Repeated measures ANOVA

3. Other Pre Specified Outcome: Net Glucose Uptake
Description: Individual net reuptake rates at each time point were calculated by the following formula: net uptake = (Cv-CA) x {FBF x [101-hematocrit/100]}, where Cv and CA represent the concentration of glucose in the brachial vein and artery, respectively.
Time Frame: At baseline and after maximum dose of bradykinin
Measure: Mean (Standard Error); unit: microgram/min/100ml
Arm/Group | Control | L-NMMA + Control | Isosorbide + L-NMMA + Control | Sildenafil + L-NMMA + Control
Number analyzed (Participants) | 24 | 23 | 11 | 12
microgram/min/100ml
  Net glucose uptake (bradykinin 0 ng/min) | -79.95 (22.894) | -74.36 (7.125) | -71.4 (27.74) | -67.3 (13.17)
  Net glucose uptake (bradykinin 200 ng/min) | -319.85 (97.109) | -142.86 (49.935) | -163.233 (36.504) | -125.32 (45.705)

ADVERSE EVENTS:
Arm/Group | All Participants
Serious Adverse Events (participants affected / at risk) | 0/24
Other Adverse Events (participants affected / at risk) | 4/24
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants (N=24)
Headache (Nervous system disorders) | 2 (2)
fainted (Nervous system disorders) | 1 (1)
unexpected drug response (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No